CLINICAL TRIAL: NCT07367256
Title: Efficacy of a Virtual Reality-Mediated Intervention on Emotion Recognition and Understanding in Children With Autism Spectrum Disorder
Brief Title: Using Virtual Reality to Improve Emotion Understanding in Children With Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto per la Ricerca e l'Innovazione Biomedica (Other)
Responsible Party: Principal Investigator, Flavia Marino, Head of Unit, Istituto per la Ricerca e l'Innovazione Biomedica
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CNR-IRIB-PRO-2026-002
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Autism; Autism Disorder
Keywords: autism; children; emotional skills; virtual reality; emotional recognition
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group with virtual reality (Experimental): The intervention protocol is designed to enhance socio-emotional skills in children with high-functioning autism spectrum disorder. The intervention focuses on the recognition and understanding of basic and complex emotions, the expansion of emotional vocabulary, and the ability to associate situations, thoughts, and emotions, promoting the differentiation between mental and emotional states.
  The treatment consists of weekly sessions over a total duration of four months and is structured around gradual activities based on visual stimuli and everyday social situations. These activities are carried out by the experimental group through the use of immersive virtual reality technology (Oculus), which allows children to interact with structured environments and scenarios designed to facilitate emotional and social learning.
  Interventions: Other: Oculus intervention
- Control group (Other): The control group follows the same intervention protocol aimed at enhancing socio-emotional skills in children with high-functioning autism spectrum disorder. In this group as well, the intervention focuses on the recognition and understanding of basic and complex emotions, the expansion of emotional vocabulary, and the ability to associate situations, thoughts, and emotions, promoting the differentiation between mental and emotional states.
  The treatment consists of weekly sessions over a total duration of four months and is structured around gradual activities based on visual stimuli and everyday social situations. However, unlike the experimental group, the activities are conducted in a traditional format, without the use of immersive technology (Oculus), with the therapist directly guiding the child through the activities and supporting their emotional and social understanding.
  Interventions: Other: Traditional intervention

INTERVENTIONS:
Other: Oculus intervention — Phase 1: Basic Emotions (happiness, sadness, anger, fear, disgust, surprise)
  * Step 1-3: Sequential recognition and identification of emotions on faces, using sets of 4 or 6 images.
  * Step 4-6: Association of thoughts, emotions, and situations in everyday scenarios.
  All activities are conducted through immersive virtual reality (Oculus), allowing children to interact with structured environments and scenarios that facilitate socio-emotional learning.
  Phase 2: Complex Emotions (guilt, shame, pride, frustration, jealousy)
  * Step 1-6: Same structure as Phase 1, using complex emotions.
  * Activities are mediated via Oculus, providing an interactive and immersive learning experience
  Arms: Experimental group with virtual reality
Other: Traditional intervention — Phase 1: Basic Emotions (happiness, sadness, anger, fear, disgust, surprise)
  * Step 1-3: Sequential recognition and identification of emotions on faces, using sets of 4 or 6 images.
  * Step 4-6: Association of thoughts, emotions, and situations in everyday scenarios.
  All activities are conducted in a traditional format, without the use of immersive technology, with the therapist guiding the child directly through the exercises to support socio-emotional learning.
  Phase 2: Complex Emotions (guilt, shame, pride, frustration, jealousy)
  * Step 1-6: Same structure as Phase 1, using complex emotions.
  * Activities are performed under direct therapist supervision in a non-technological setting.
  Arms: Control group

SUMMARY:
Autism Spectrum Disorders (ASD) are neurodevelopmental conditions characterized by difficulties in social interaction, communication, and in understanding one's own and others' mental and emotional states. In particular, skills related to the recognition, understanding, and regulation of emotions represent a significant area of vulnerability in children with high-functioning ASD, with important consequences for social and relational functioning.

The present study aims to evaluate the effectiveness of an intervention protocol designed to enhance socio-emotional understanding, with a specific focus on the recognition of basic and complex emotions, the expansion of emotional vocabulary, the association between situations, thoughts, and emotions, and the differentiation between thoughts and emotions. Furthermore, the study seeks to investigate the role of immersive technology (Oculus) as a potential facilitator of emotional learning compared to a traditional intervention approach. The sample will consist of children with a diagnosis of high-functioning ASD, aged between 7 and 10 years, with sentence-level language abilities, the capacity to narrate non-present events, and an intellectual quotient above 80 (assessed using the Griffiths Scales or the WISC-IV). Participants will be divided into two groups: an experimental group (OCULUS), which will receive the intervention mediated by the use of Oculus technology, and a control group which will undergo the same protocol without technological support.

ELIGIBILITY:
Inclusion Criteria:

* Language in sentences
* Ability to narrate events not present
* QS/QI>80

Exclusion Criteria:

* presence of other medical disorders

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Test of Emotional Vocabulary (TLE) | The administration has a duration of 15 minutes.
  The test contains an initial board, with which the child is introduced to the two protagonists of the subsequent stories, a boy and a girl; there is then a pretest board and 14 storyboards. For each of them, the examiner reads the short story to the child and then asks the child to choose, from two alternative emotional words, the one that best expresses what the protagonist of the story is feeling. In the first part, the child's understanding of emotional vocabulary referring to six basic emotions plus one complex emotion (joy, happiness, sadness, anger, fear, disgust and shame) is assessed; in the second part, the emotional terms all refer to complex emotions (guilt, envy, jealousy, contempt, hate, longing and pride).

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Marino, Principal Investigator — Institute for Biomedical Research and Innovation (IRIB) - National Research Council (CNR)
Locations (1):
- Istituto per la Ricerca e l'Innovazione Biomedica, Messina, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Papoutsi, C., Drigas, A., & Skianis, C. (2021). Virtual and augmented reality for developing emotional intelligence skills. Int. J. Recent Contrib. Eng. Sci. IT (IJES), 9(3), 35-53.
- [Background] Frolli A, Savarese G, Di Carmine F, Bosco A, Saviano E, Rega A, Carotenuto M, Ricci MC. Children on the Autism Spectrum and the Use of Virtual Reality for Supporting Social Skills. Children (Basel). 2022 Feb 1;9(2):181. doi: 10.3390/children9020181. PMID 35204903
- [Background] American Psychiatric Association. (2013). Diagnostic and statistical manual of mental disorders (5th ed.) https://doi.org/10.1176/appi.books.9780890425596.